CLINICAL TRIAL: NCT06591884
Title: Evaluation of the Efficacy of 0.08% Tacrolimus Nanoencapsulated Aqueous Solution Spray Vs. 0.1% Free Tacrolimus Commercial Ointment in the Treatment of Oral Lichen Planus - a Randomized Clinical Trial
Brief Title: Evaluation of the Efficacy of 0.08% Tacrolimus Nanoencapsulated Aqueous Solution Spray Vs. 0.1% Free Tacrolimus Commercial Ointment in the Treatment of Oral Lichen Planus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0566; 76823524.3.1001.5327 (Other: Hospital de Clinicas de Porto Alegre)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Oral Erosive Lichen Planus
Keywords: Oral Lichen Planus; Tacrolimus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.08% tacrolimus nanoencapsulated aqueous solution spray (Experimental): tacrolimus modified-release
  Interventions: Drug: Tacrolimus modified-release
- 0.1% free tacrolimus commercial ointment (Active Comparator)
  Interventions: Drug: tacrolimus ointment 0.1%

INTERVENTIONS:
Drug: Tacrolimus modified-release — 0.08% tacrolimus nanoencapsulated aqueous solution spray
  Arms: 0.08% tacrolimus nanoencapsulated aqueous solution spray
Drug: tacrolimus ointment 0.1% — 0.1% free tacrolimus commercial ointment
  Arms: 0.1% free tacrolimus commercial ointment

SUMMARY:
The goal of this clinical trial is to assess the efficacy of different formulations of the drug tacrolimus in treating patients with oral lichen planus. The main questions it aims to answer are:

* Does the nanoencapsulation of tacrolimus in an aqueous solution, used as a spray, improve the effectiveness of treating oral lichen planus lesions compared to the commercially available tacrolimus ointment?
* Which tacrolimus formulation can keep participants free of lesions for longer periods?

Researchers will compare a spray of 0.08% tacrolimus nanoencapsulated aqueous solution against a 0.1% free tacrolimus commercial ointment to determine which formulation is more effective.

Participants will:

* Apply one of the proposed tacrolimus formulations twice a day for 1 month.
* Visit the clinic once every 2 weeks for checkups and tests, with follow-ups extending up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a clinical and histopathological diagnosis of erosive/ulcerative/atrophic and symptomatic oral lichen planus, according to the criteria established by the American Academy of Oral and Maxillofacial Pathology

Exclusion Criteria:

* History of oral cancer;
* history of allergic reactions to tacrolimus or any other component of the formulas;
* history of organ transplant or have a systemic condition that induces significant immunosuppression;
* be pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Oral Disease Severity Score (ODSS) - 50% | 30 days
  Number of patients achieving a reduction of at least 50% in ODSS score compared to baseline and the percentage and absolute reduction in ODSS score in both groups at the end of treatment (30 days).
  ODSS score ranges from 0 to 106, lower score mean a better outcome.
VAS (visual analogical score) pain score - 50% | 30 days
  number of patients achieving a reduction of at least 50% in VAS score of reported pain compared to baseline and the percentage and absolute reduction in VAS score in both groups at the end of treatment (30 days).
  VAS score ranges from 0 to 10, lower score mean a better outcome.

SECONDARY OUTCOMES:
OHIP-14 quality of life score | 15-90 days
  the percentage and absolute reduction in OHIP-14 scale score in both groups at mid-treatment and end of treatment (15 and 30 days) and at the 30 and 60-day follow-ups after treatment completion (follow-up 1 and follow-up 2).
  OHIP-14 score ranges from 0 to 56, lower score mean a better outcome.
Beck scale scores (anxiety levels) | 15-90 days
  The percentage and absolute reduction in Beck scale score in both groups at mid-treatment and end of treatment (15 and 30 days) and at the 30 and 60-day follow-ups after treatment completion (follow-up 1 and follow-up 2).
  OHIP-14 score ranges from 0 to 63, lower score mean a better outcome.
hedonic scale satisfaction scores | 30-90 days
  Comparison of hedonic scale scores of satisfaction reported by the participants in regards of treatment received in both groups at the end of treatment (30 days) and at the 30 and 60-day follow-ups after treatment completion (follow-up 1 and follow-up 2).
  Hedonic scale satisfaction score ranges from 0 to 9, higher score mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Visioli, DDS, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No